CLINICAL TRIAL: NCT01946126
Title: A Retrospective Chart Review to Evaluate Diagnosis and Treatment of Chronic Migraine and Headache
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-BTX-CM-13-592
Record Dates: First submitted 2013-09-17; First posted 2013-09-19 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Migraine Disorders; Headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Migraine Diagnosis: This is a retrospective chart review for patients diagnosed with Chronic Migraine. There is no intervention in this study.
  Interventions: Other: No Intervention
- Other Headache Diagnoses: This is a retrospective chart review of patients with headache diagnoses other than Chronic Migraine. There is no intervention in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention in this study.

SUMMARY:
This study is a retrospective chart review in patients diagnosed with headache or migraine to evaluate treatment patterns and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic migraine or other diagnosis of migraine or headache for a minimum of 15 months
* Eight (8) headache days per month for at least 1 of the preceding 15 months

Exclusion Criteria:

* Not currently diagnosed with chronic migraine, headache or migraine
* History of receiving botulinum toxin injections for the treatment of chronic migraine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of chronic migraine or other diagnosis of migraine or headache.
Sampling Method: Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Raleigh, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Migraine Diagnosis | Other Headache Diagnoses
Started | 184 | 275
Completed | 184 | 275
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Migraine Diagnosis | Other Headache Diagnoses | Total
Number analyzed (Participants) | 184 | 275 | 459
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.02 (11.54) | 45.44 (11.62) | 45.3 (11.58)
Sex/Gender, Customized [Number; unit: Participants] | NA — Gender was not collected in this study. | NA — Gender was not collected in this study. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Presence or Absence of Prophylactic Medication for Headache/Migraine
Description: The presence or absence of prophylactic medications used by the subject for headache/migraine is evaluated through the study period.
Time Frame: 15 Months
Population: All enrolled subjects
Measure: Number; unit: Participants
Arm/Group | Chronic Migraine Diagnosis | Other Headache Diagnoses
Number analyzed (Participants) | 184 | 275
Participants
  Presence of Prophylactic Medication | 166 | 227
  Absence of Prophylactic Medication | 18 | 48

2. Secondary Outcome: Number of Unique Prophylactic Medications for Headache/Migraine Reported
Description: The numbers of unique prophylactic medications used by the subjects for headache/migraine are evaluated through the study period.
Time Frame: 15 Months
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: Medications
Arm/Group | Chronic Migraine Diagnosis | Other Headache Diagnoses
Number analyzed (Participants) | 184 | 275
Medications | 2.7 (1.49) | 1.8 (1.27)

3. Secondary Outcome: Number of Days With a Headache Recorded at the Visit With the Highest Number of Headaches
Description: The number of headache days is reported at the visit with the highest number of headaches.
Time Frame: 15 Months
Population: All enrolled subjects
Measure: Mean (95% Confidence Interval); unit: Headache Days
Arm/Group | Chronic Migraine Diagnosis | Other Headache Diagnoses
Number analyzed (Participants) | 184 | 275
Headache Days | 22.0 [20.6 to 23.4] | 19.2 [18.2 to 20.2]

4. Secondary Outcome: Highest Number of Headache Days Per Month at a Qualifying Visit
Description: The highest number of headache days per month are reported at a qualifying visit per the medical record.
Time Frame: 15 Months
Population: All enrolled subjects with data for this outcome measure
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Chronic Migraine Diagnosis | Other Headache Diagnoses
Number analyzed (Participants) | 133 | 183
Days | 16.28 [14.4 to 18.2] | 14.01 [12.6 to 15.4]

5. Secondary Outcome: Number of Visits for Headache Diagnosis
Description: The number of visits for headache diagnosis is evaluated through the study period.
Time Frame: 15 Months
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Chronic Migraine Diagnosis | Other Headache Diagnoses
Number analyzed (Participants) | 184 | 275
Visits | 4.7 (2.5) | 3.5 (1.63)

ADVERSE EVENTS:
Description: Adverse events (AEs) and serious adverse events (SAEs) were not collected in this study.
Arm/Group | Chronic Migraine Diagnosis | Other Headache Diagnoses
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.